CLINICAL TRIAL: NCT00456001
Title: Study to Compare the Heparin Induced Thrombocytopenia Rates Associated With Heparin and Low Molecular Weight Heparin Usage as Well as Evaluate the Economic and Long-Term Clinical Burden of Heparin Induced Thrombocytopenia.
Brief Title: Heparin Induced Thrombocytopenia: Pharmacoeconomics
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Samuel Z. Goldhaber, MD, Brigham and Women's Hospital
Other Study IDs: 2006-P-001982
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: Heparin Induced Thrombocytopenia (HIT)
Keywords: heparin; low molecular weight heparin; enoxaparin; anticoagulation; thrombosis; venous thrombosis; thromboembolism; pulmonary embolism; medication
MeSH Terms: conditions — Thrombosis; Venous Thrombosis; Thromboembolism; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients at BWH receiving unfractionated heparin or enoxaparin who subsequently develop heparin induced thrombocytopenia will be identified via a computer generated report designed for the purposes of this study.

Subsequently, we will compare the heparin induced thrombocytopenia rates associated with heparin and low molecular weight heparin usage as well as evaluate the economic and long-term clinical burden of heparin induced thrombocytopenia.

DETAILED DESCRIPTION:
The goal of this research is to investigate the outcomes and pharmacoeconomics of patients diagnosed with heparin induced thrombocytopenia (HIT).

Background:

Heparin induced thrombocytopenia (HIT) is a complication of heparin therapy receiving wide-scale awareness, increasing detection, and concern. Data from controlled studies demonstrate a lower incidence of HIT with low molecular-weight heparin (LMWH) when compared to unfractionated heparin (UFH) However, registry data comparing the incidence of HIT in patients receiving LWMH vs. UFH are scarce. We will define the incidence of HIT in patients receiving LWMH vs. UFH in the "real world" setting at Brigham and Women's Hospital. We will evaluate the associated clinical and economic implications.

Our Objectives are:

1. Compare the HIT rates associated with heparin and LMWH usage:

   The incidence of HIT will be assessed for initial the type of heparin exposure responsible for causing HIT. Patients will be categorized as receiving UFH with or without LMWH or as receiving only LMWH.
2. Evaluate the economic burden of HIT to hospitals and/or payors:

   We will capture all expenses associated with each patient admission. Hospital expenses will be tabulated daily using the hospital database and the proprietary cost accounting system, Transition Systems, Inc (TSI).

   Expenses will be categorized by procedure or area of care and will include Emergency Department care, operating room use, hospital room and board, hospital based physician fees, nursing labor, dialysis, clinical laboratory studies (hematology, microbiology, cytology, urinalysis), radiology (magnetic resonance imaging, computer axial tomography, and ultrasound imaging), ancillary services (support nutrition support, occupational, respiratory, and physical therapy services), medications, diagnostic procedures (cardiac catheterization, electrophysiologic testing, endoscopy, vascular ultrasound, pathology), and diagnostic testing (electrocardiogram, electroencephalogram, and electromyography).

   We will compare the mean total hospitalization costs of UFH induced HIT to those associated with LMWH induced HIT. Where possible we will compare individual resources used within the two groups.
3. Evaluate the long-term clinical burden and recurrence of HIT:

All patients diagnosed with HIT during the study period will be evaluated for a documented prior diagnosis of HIT. Additionally, all patients will be monitored for 12 months following initial diagnosis of HIT for subsequent diagnosis of HIT. The long-term clinical burden of HIT will be assessed by tracking the rates of in-hospital and subsequent mortality.

Patient Identification:

Brigham and Women's Hospital has a sophisticated computerized system that integrates medical, laboratory, and pharmacy data. Patients receiving UFH or enoxaparin who subsequently develop HIT will be identified via a computer generated report designed for the purposes of this study.

All patients with a diagnosis of HIT during the study period (January 2004 - December 2005) will be included in the evaluation. Criteria for a HIT positive diagnosis include: a clinical suspicion of HIT, a decrease in platelets to <150,000 or 50% from baseline, and serologic confirmation defined as a positive PF4 ELISA test. Patients will be monitored for clinical symptoms of HIT (new thrombosis, thrombocytopenia). Patients will be followed for clinical outcomes and incurred expenses over the hospitalization period and subsequent outpatient follow up.

Data Collection:

A protocol specific database will be created on an Access platform to house all collected data. Data will be analyzed internally by the Venous Thromboembolism Research Group.

ELIGIBILITY:
All patients hospitalized at BWH who have a PF4-Positive antibody test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients hospitalized at BWH who have a PF4-Positive antibody test
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Clotting and Bleeding Complications | 90 Days

SECONDARY OUTCOMES:
Mortality | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z. Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Baroletti SA, Goldhaber SZ. Heparin-induced thrombocytopenia. Circulation. 2006 Aug 22;114(8):e355-6. doi: 10.1161/CIRCULATIONAHA.106.632653. No abstract available. PMID 16923760
- See also: North American Thrombosis Forum — http://www.NATFonline.org